CLINICAL TRIAL: NCT02190552
Title: A.R.I.S.E. Analysis of Revascularisation in Ischemic Stroke With EmboTrap: Post Marketing Observational Study of CE Marked EmboTrap Mechanical Thrombectomy Device
Brief Title: Analysis of Revascularisation in Ischemic Stroke With EmboTrap
Acronym: ARISE
Status: Terminated | Type: Observational
Sponsor: Neuravi Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP001
Record Dates: First submitted 2014-07-10; First posted 2014-07-15 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2018-11

CONDITIONS: Ischemic Stroke
Keywords: Brain; Brain Clot; Brain Diseases; Brain Infarction; Cerebral Ischemia; Cerebrovascular Disorders; EmboTrap® Revascularization Device; EmboTrap; Ischemia; Ischemic; Ischemic Stroke; Mechanical Thrombectomy; Neurovascular Intervention; Revascularization; Stent Retriever; Stroke; Vascular Diseases
MeSH Terms: conditions — Ischemic Stroke; Brain Diseases; Brain Infarction; Brain Ischemia; Cerebrovascular Disorders; Ischemia; Stroke; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- EmboTrap® Revascularization Device: The EmboTrap® Revascularization Device is the investigational device
  Interventions: Device: EmboTrap® Revascularization Device

INTERVENTIONS:
Device: EmboTrap® Revascularization Device
  Other Names: EmboTrap

SUMMARY:
A.R.I.S.E. is a post approval observational study using standard care. The purpose of this study is to collect information about the ability of the EmboTrap device to remove blood clots from the brain, and the associated performance characteristics and clinical outcomes. No formal hypothesis testing is needed as no comparisons are planned within the study. Instead, estimates of each population parameter of interest for all primary and secondary endpoints will be provided using appropriate confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* The patient or the patient's legally authorized representative has signed and dated an Informed Consent Form.
* Aged between 18 years and 80 years (inclusive).
* A new focal disabling neurologic deficit consistent with acute cerebral ischemia.
* NIHSS score ≥8 and ≤25.
* Pre-ictal mRS score of 0 or 1.
* Angiographic confirmation of an occlusion of an ICA (including T and L occlusions), M1 or M2, MCA, or BA with TICI flow of 0-1.
* Confirmation by the interventionalist, after screening CT or MRI, that the treatment site can be accessed with the Neuravi device.
* The interventionalist estimates that at least one deployment of the Neuravi device can be completed within 5 hours from the onset of symptoms, or if time of onset of symptoms is unknown or > 5 hours, patients can be included using imaging with the following criteria:

  1. MRI criterion: ASPECTS 8 to 10, or,volume of diffusion restriction ≤30 mL and mismatch between perfusion reduction and diffusion restriction present.
  2. CT criterion: ASPECTS 8 to 10 on baseline CT or CTA-source images, or, volume of significantly lowered CBV ≤30 mL and mismatch between perfusion reduction and low CBV present.

Exclusion Criteria:

* Life expectancy of less than 6 months.
* Females who are pregnant or lactating.
* History of severe allergy to contrast medium.
* Has suffered a stroke in the past three months.
* The patient presents with an NIHSS score <8 or >25 or is physician assessed as being in a clinically relevant uninterrupted coma.
* Use of warfarin anticoagulation with International Normalized Ratio (INR) > 3.0.
* Platelet count < 50,000.
* Glucose < 50 mg/dL.
* Heparin use in previous 24 hours with PTT or ACT > 2X normal.
* Any known hemorrhagic or coagulation deficiency.
* Computed tomography (CT) or Magnetic Resonance Imaging (MRI) evidence of recent/ fresh hemorrhage on presentation.
* For basilar artery occlusion, extended early ischemic changes as confirmed by pc-ASPECTS ≤ 7 on baseline CT or CTA-source images, or extensive DWI lesions in the midbrain or pons regions on pre-treatment MRI.
* Baseline CT or MRI showing mass effect or intracranial tumor (except small meningioma).
* Excessive arterial tortuosity that precludes the study device from reaching the target vessel.
* A proximal stenosis or complete occlusion that cannot, as judged by the responsible interventionalist, be treated safely or which prevents access to the occluded vessel with the Neuravi device.
* Evidence of active infection.
* Known cancer with metastases
* Current use of cocaine or other vasoactive substance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ischemic stroke patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Tommy Andersson, Principal Investigator — Karolinska Institutet; Prof. Dr. Heinrich Mattle, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (5):
- Aarhus University Hospital, Aarhus, Denmark
- Universitätsklinikum Kiel, Kiel, Germany
- Beaumont Hospital, Dublin, Ireland
- Hospital Clinico de Barcelona, Barcelona, Spain
- Karolinska Institutet, Solna, Sweden

REFERENCES:
- [Derived] Mattle HP, Scarrott C, Claffey M, Thornton J, Macho J, Riedel C, Soderman M, Bonafe A, Piotin M, Newell J, Andersson T; ARISE I Study Group. Analysis of revascularisation in ischaemic stroke with EmboTrap (ARISE I study) and meta-analysis of thrombectomy. Interv Neuroradiol. 2019 Jun;25(3):261-270. doi: 10.1177/1591019918817406. Epub 2018 Dec 18. PMID 30563388
- See also: Company website — http://neuravi.com

RESULTS

PARTICIPANT FLOW:
Groups:
- EmboTrap® Revascularization Device: The EmboTrap® Revascularization Device is the investigational device
  EmboTrap® Revascularization Device
Period: Overall Study
Arm/Group | EmboTrap® Revascularization Device
Started | 40
Completed | 36
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | EmboTrap® Revascularization Device
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 14
  Ireland | 4
  Germany | 6
  Spain | 10
  France | 6
National Institutes of Health Stroke Scale (NIHSS) Score [Mean (Standard Deviation); unit: units on a scale] — The NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. NIHSS scores range from 0 - 42. A score of 0 indicates no stroke symptoms. Higher scores indicate incremental levels of neurological impairment.
  units on a scale | 15 (5)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27 (4)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Revascularisation Following the Use of the Neuravi Device.
Description: Revascularisation is defined as achieving a modified Thrombolysis in Cerebrovascular Infarction (mTICI) score of 2b or greater.
  mTICI is a 6-point grading system for determining the response of thrombolytic therapy for ischaemic stroke:
  mTICI 0 = No perfusion
  mTICI 1 = Penetration but not perfusion
  mTICI 2a = Some perfusion with distal branch filling of <50% of territory visualized
  mTICI 2b = Substantial perfusion with distal branch filling of ≥50% of territory visualized
  mTICI 2c = Near-complete perfusion
  mTICI 3 = Complete perfusion
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | EmboTrap® Revascularization Device
Number analyzed (Participants) | 39
Participants | 28

2. Secondary Outcome: Time to Revascularization
Description: Defined as time from groin puncture to visualization of final angiographic result.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | EmboTrap® Revascularization Device
Number analyzed (Participants) | 39
minutes | 76 (50)

3. Secondary Outcome: Mortality Post Procedure
Description: All procedure related mortality (i.e. directly traceable to a procedure related SAE).
Time Frame: 7 and 90(±14) days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | EmboTrap® Revascularization Device
Number analyzed (Participants) | 40
Participants
  Procedure-related Mortality at Day 7 | 0
  All cause Mortality at Day 90 | 4

4. Secondary Outcome: Serious Adverse Device Related Effects (SADE)
Description: SADE is defined as vessel perforation or vessel dissection, which is attributable to the Neuravi device, or where the Neuravi device cannot be ruled out as the cause.
Time Frame: 24(-8/+12) hours Post Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | EmboTrap® Revascularization Device
Number analyzed (Participants) | 40
Participants | 0

5. Secondary Outcome: Symptomatic ICH
Description: Symptomatic ICH rate within 24 hours (range: 16 to 36 hours) post-procedure. Symptomatic intracranial haemorrhage (parenchymatous haemorrhage type 2), at post-treatment scan combined with neurological deterioration (C2) leading to an increase of 4 points or more on the NIH Stroke Scale.
  The NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. NIHSS scores range from 0 - 42. A score of 0 indicates no stroke symptoms. Higher scores indicate incremental levels of neurological impairment.
Time Frame: 24(-8/+12) hours Post Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | EmboTrap® Revascularization Device
Number analyzed (Participants) | 40
Participants | 0

6. Secondary Outcome: Clinical Outcome at 90 Days
Description: A good clinical outcome will be judged to be a mRS score of ≤2 at 90(±14) days.
  mRS is a scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. mRS scores range from 0 to 6:
  mRS 0 = No symptoms.
  mRS 1 = No significant disability.
  mRS 2 = Slight disability.
  mRS 3 = Moderate disability.
  mRS 4 = Moderately severe disability.
  mRS 5 = Severe disability.
  mRS 6 = Dead.
Time Frame: 90(±14) days Post Procedure
Population: Data was not collected for all participants.
Measure: Count of Participants; unit: Participants
Arm/Group | EmboTrap® Revascularization Device
Number analyzed (Participants) | 30
Participants | 20

7. Secondary Outcome: Rate of New Territory Embolization
Description: Embolization, or thrombus dislocation, into a previously uninvolved vascular territory as evaluated from angiographic images by the Angiography Core Lab and the Data Safety Monitoring Board.
Time Frame: 24(-8/+12) hours Post Procedure
Population: Data were not collected
Arm/Group | EmboTrap® Revascularization Device
Number analyzed (Participants) | 0

8. Secondary Outcome: Evidence of Infarction
Description: Infarction, of a previously uninvolved vascular territory, as evaluated from 24hr Computed Tomography imaging by the Angiography Core lab.
Time Frame: 24(-8/+12) hours Post Procedure
Population: Data were not collected
Arm/Group | EmboTrap® Revascularization Device
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | EmboTrap® Revascularization Device
Serious Adverse Events (participants affected / at risk) | 9/40
Other Adverse Events (participants affected / at risk) | 24/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EmboTrap® Revascularization Device (N=40)
Pneumonia (Infections and infestations) | 1
Stroke in evolution (Nervous system disorders) | 4
Embolism (Nervous system disorders) | 1
Neurological Deterioration (Nervous system disorders) | 1
Occlusion (Nervous system disorders) | 1
Pseudoaneurysm (Vascular disorders) | 1
Vessel perforation (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EmboTrap® Revascularization Device (N=40)
Atrial Fibrillation (Cardiac disorders) | 2
Bradycardia (Cardiac disorders) | 3
Other Cardiac disorders (Cardiac disorders) | 2
Pneumonia (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 5
Blood potassium decreased (Investigations) | 2
Embolism (Nervous system disorders) | 2
Haemorrhagic transformation stroke (Nervous system disorders) | 2
Other Respiratory disorders (Respiratory, thoracic and mediastinal disorders) | 2
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No